CLINICAL TRIAL: NCT00904124
Title: Determination of the Effect of Different Types of Isolated Dietary Fiber on ad Libitum Food Intake in Healthy Human Subjects
Brief Title: The Effect of Different Types of Dietary Fiber on Satiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Prof. Dr. E. Feskens, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 0902-face
Record Dates: First submitted 2009-05-17; First posted 2009-05-19 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
Keywords: Dietary fiber; guar gum; alginate; cellulose; food intake; eating behaviour
MeSH Terms: conditions — Feeding Behavior | interventions — Cellulose; Alginates; guar gum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Control (Placebo Comparator): No regular flour replaced
  Interventions: Dietary Supplement: cellulose, alginate, guar gum
- 5% Cellulose (Experimental): 5% regular flour is replaced by cellulose
  Interventions: Dietary Supplement: cellulose, alginate, guar gum
- 2.5% Alginate (Experimental): 2.5% regular flour is replaced by Alginate
  Interventions: Dietary Supplement: cellulose, alginate, guar gum
- 5% Alginate (Experimental): 5% regular flour is replaced by Alginate
  Interventions: Dietary Supplement: cellulose, alginate, guar gum
- 2.5% Guar gum (Experimental): 2.5% regular flour is replaced by Guar gum
  Interventions: Dietary Supplement: cellulose, alginate, guar gum
- 1.25% Guar gum (Experimental): 1.25% regular flour is replaced by Guar gum
  Interventions: Dietary Supplement: cellulose, alginate, guar gum

INTERVENTIONS:
Dietary Supplement: cellulose, alginate, guar gum — 6 different food products are developed with different dosages of dietary fiber. Regular flour is replaced by dietary fiber, dosages are described in the 'arms'section.

SUMMARY:
It has been suggested that dietary fibers can affect food intake and satiation. Satiation, or meal termination, can be induced by sensory properties and energy density of fiber-rich food products, but also by the chemical/physical/rheological behavior of the fibers in the stomach and/or intestine. It is not clear which properties are the key regulators of satiation by fiber sources. There are many types of dietary fiber, which have diverse sensory and chemical properties, thus these might have different effects on satiation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-50 years
* BMI: 18-25 kg/m2
* Healthy: as judged by the participant

Exclusion Criteria:

* Weight loss or weight gain of more than 5 kg during the last 2 months
* Using an energy restricted diet during the last 2 months
* Lack of appetite for any (unknown) reason
* Having problems with chewing and swallowing
* Having problems with digestion
* Restrained eater
* Hypersensitivity for gluten or other ingredients of chocolate cookies
* Hypersensitivity for one of the fibers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Ad libitum intake | 1 hour and 2 hours

SECONDARY OUTCOMES:
eating rate | 1 hour and 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Edith Feskens, Dr, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands

REFERENCES:
- [Derived] Wanders AJ, Jonathan MC, van den Borne JJ, Mars M, Schols HA, Feskens EJ, de Graaf C. The effects of bulking, viscous and gel-forming dietary fibres on satiation. Br J Nutr. 2013 Apr 14;109(7):1330-7. doi: 10.1017/S0007114512003145. Epub 2012 Jul 31. PMID 22850326